CLINICAL TRIAL: NCT03551834
Title: Ahmed Glaucoma Valve Implantation; Graft-Free Short Tunnel Small Flap Versus Scleral Patch Graft
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shahid Beheshti University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Zahra Rabbani Khah, Clinical Professor, Shahid Beheshti University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 97122
Record Dates: First submitted 2018-05-16; First posted 2018-06-11 (Actual); Last update posted 2018-06-11 (Actual); Status verified 2018-05

CONDITIONS: Glaucoma
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- doing scleral patch graft glaucoma implantation (Active Comparator)
  Interventions: Other: Conventional scleral patch graft glaucoma implantation
- Using short tunnel small flap technique (Active Comparator)
  Interventions: Other: New surgical method (short tunnel small flap technique)

INTERVENTIONS:
Other: Conventional scleral patch graft glaucoma implantation — conventional AGV implantation by using scleral patch graft to cover the tube and prevent tube exposure
  Arms: doing scleral patch graft glaucoma implantation
Other: New surgical method (short tunnel small flap technique) — a novel technique named short tunnel small flap (STSF) by tunneling the sclera to pass the AGV tube without using scleral patch graft.
  Arms: Using short tunnel small flap technique

SUMMARY:
Glaucoma implants have been used for refractory glaucoma and are gaining popularity as a primary procedure in selected patients. In order to prevent tube erosion, a biologic material such as pericardium, cornea, and sclera is used as coverage over the tube. Despite this preventive measures, patch graft thinning and silicon tube exposure are still a serious complications and may occur in 1%-7% of eyes after glaucoma implantation. In this study we used a novel technique named short tunnel small flap (STSF) by tunneling the sclera without using any biological material . efficacy and safety of this technique is comparing with conventional scleral patch graft.

This randomized clinical trial, was performed at the Glaucoma Clinic of Labbafinejad Medical Center, Tehran, IRAN from September 2015 to January 2017 . The study was approved by the ethics committee at the Ophthalmic Research Center, Shahid Beheshti University of Medical Sciences, Tehran, Iran and followed the tenets of the Declaration of Helsinki. After explaining all therapeutic options and their side effects, the written consent form was obtained from all patient. 80 eyes of 80 patients with refractory glaucoma underwent AGV implantation by short tunnel small flap technique (group1) or scleral patch graft (group2) randomly. Primary outcome measure is Intraocular pressure(IOP) and Tube exposure, and secondary outcome measure is success rate that is defined as intraocular pressure (IOP) > 5 mmHg, ≤ 21 mmHg, and IOP reduction ≥ 20% from baseline at two consecutive visits after three months, no reoperation for glaucoma. Outcome measures are compared at 1, 3 , 6 and 12 months postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* Iranian patients with Caucasian ethnicity, and at least 25 years old who had inadequately controlled glaucoma.

Exclusion Criteria:

* Primary congenital glaucoma, thin sclera, no light perception vision, pregnant or nursing women, iridocorneal endothelial syndrome, epithelial or fibrous down growth, and unwillingness to participate in the study.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2017-01-20 (Actual); Primary Completion 2017-09-20 (Actual); Study Completion 2018-09 (Estimated)

PRIMARY OUTCOMES:
Intraocular pressure(IOP) | 12 months post operatively
  Goldmann applanation tonometry
Tube exposure | 12 months post operatively
  slit lamp examination

SECONDARY OUTCOMES:
success rate | 12 months
  Success rate defined as intraocular pressure (IOP) > 5 mmHg, ≤ 21 mmHg, and IOP reduction ≥ 20% from baseline at two consecutive visits after three months, no reoperation for glaucoma

CONTACTS AND LOCATIONS:
Locations (1):
- Ophthalmic Research Center, Tehran, Iran